CLINICAL TRIAL: NCT04401527
Title: Treatment of Lung Injury From COVID-19 Infection With Intravenous Sodium Nitrite: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Clinical Study
Brief Title: Treatment of Lung Injury From COVID-19 Infection With Intravenous Sodium Nitrite
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Hope Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SN02-01
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; Acute Respiratory Failure
Keywords: COVID-19; Acute Respiratory Distress Syndrome; Acute Respiratory Failure; ARDS; Respiratory Failure; Intubation; Mechanical Ventilation; Intubated; Mechanical Ventilator; ECMO; Sodium Nitrite; Nitrite; Nitric Oxide
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Sodium Nitrite; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Nitrite (Active Comparator): Hope Pharmaceuticals' Sodium Nitrite Injection administered by continuous intravenous infusion.
  Interventions: Drug: Sodium Nitrite
- Placebo (Placebo Comparator): 0.9% Sodium Chloride Injection, USP (normal saline) administered by continuous intravenous infusion.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Sodium Nitrite — Continuous intravenous infusion of Sodium Nitrite Injection
  Other Names: Hope Pharmaceuticals Sodium Nitrite Injection USP 30 mg/mL
  Arms: Sodium Nitrite
Drug: Normal Saline — Continuous intravenous infusion of Normal Saline
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of intravenous Sodium Nitrite Injection for treatment of patients infected with COVID-19 who develop lung injury and require mechanical ventilation.

DETAILED DESCRIPTION:
This Phase 2, multicenter, randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of intravenous Sodium Nitrite Injection for treatment of patients infected with COVID-19 who develop lung injury and require mechanical ventilation. The primary objective is to compare the two treatment groups with respect to the proportion of study subjects who are alive and free of respiratory failure at Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Diagnosed COVID-19 disease with confirmed SARS-coV-2 viral infection;
3. Able to sign the informed consent form (ICF) or next of kin/legal guardian able to sign informed consent;
4. Randomization within 24 hours of intubation and mechanical ventilation due to respiratory failure from COVID-19 infection;
5. Absolute lymphocyte count > 800 / mm3;
6. Women of childbearing potential (WCBP) must have a negative urine or serum (if anuric) pregnancy test at screening;
7. WCBP must agree to abstain from sex or use an adequate method of contraception from the time of informed consent through Day 28;
8. Males must abstain from sex with WCBP or use an adequate method of contraception from the time of informed consent through Day 28.

Exclusion Criteria:

1. Methemoglobinemia > 2%;
2. Hypotension with systemic blood pressure < 90/60 mm Hg, or uncontrolled hypotension despite vasopressor support;
3. History of sickle cell disease, thalassemia, G6PD deficiency, lung transplant, or allergy to sodium nitrite;
4. Hemoglobin < 8 gm/dL;
5. Renal impairment with creatinine clearance < 60 mL/min/1.73m2;
6. Treatment within the past 48 hours with allopurinol (a medication that could interfere with nitrite metabolism);
7. Treatment within the past 24 hours with organic nitrates such as nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, sodium nitroprusside, and inhaled nitric oxide;
8. Treatment within the past 24 hours with lidocaine, prilocaine, benzocaine, and dapsone;
9. Requiring extracorporeal membrane oxygenation (ECMO);
10. Subjects with bacterial or fungal infections except for mild cutaneous infections or sinus infections;
11. Subjects who are pregnant or lactating;
12. Any condition that, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study;
13. Clinically relevant serious co-morbid medical conditions including, but not limited to, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, uncontrolled chronic obstructive or chronic restrictive pulmonary disease, active central nervous system (CNS) disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV) (except if HIV subject has undetectable viral load and a CD4 count of ≥ 500 cells/µL), and/or active hepatitis B or C, cirrhosis, or uncontrolled psychiatric illness/social situations that would limit compliance with study requirements;
14. Treatment within 30 days or 5 half-lives of that agent (whichever is shorter) before the first study drug dose using another investigational drug. Notwithstanding, prospective subjects who receive any of the following drugs or treatments before the first study drug dose or during this study may be considered for participation in this study: (1) a commercially available, FDA-approved drug or treatment used off-label for the treatment of COVID-19, or (2) a drug or treatment that has FDA Emergency Use Authorization for the treatment of COVID-19 patients;
15. Moribund or not expected to survive 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Survival with Unassisted Breathing | Day 28
  Proportion of study subjects who are alive and free of respiratory failure at Day 28

SECONDARY OUTCOMES:
Survival without Mechanical Ventilation | Day 28
  Number of days alive without mechanical ventilation from start of study through Day 28
Survival without Intensive Care | Day 28
  Number of days alive and not in the intensive care unit from start of study through Day 28.
Survival without Hospitalization | Day 28
  Number of days alive and not in hospital from start of study through Day 28.
Survival without ECMO | Day 28
  Alive on Day 28 and no use of ECMO therapy any time between start of study and Day 28.
Survival | Day 28
  Alive on Day 28

OTHER OUTCOMES:
Lung Status | Day 14
  Oxygenation index (PaO2/FIO2) at Day 14
Kidney Status (1) | Day 14
  Blood urea nitrogen (BUN) at Day 14
Kidney Status (2) | Day 14
  Creatinine at Day 14
Liver Status | Day 14
  Liver function tests (ALT and AST) at Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Hope Pharmaceuticals Medical Director, Study Director — Hope Pharmaceuticals
Locations (2):
- United States (2):
  - Participating Research Facility, Tampa, Florida
  - Participating Research Facility, Fort Worth, Texas